CLINICAL TRIAL: NCT00466960
Title: A Phase II Trial of Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) With Weekly Protein Bound Paclitaxel (Abraxane™) as Chemoimmunotherapy for Platinum-Refractory/Resistant Epithelial Ovarian, Primary Peritoneal and Fallopian Tube Cancer
Brief Title: Sargramostim and Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Advanced Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer That Did Not Respond to Previous Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Goff, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6168; NCI-2010-00556 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Brenner Tumor; Fallopian Tube Cancer; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mixed Epithelial Carcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Undifferentiated Adenocarcinoma; Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (colony stimulating factor and chemotherapy) (Experimental): INDUCTION THERAPY: Patients receive GM-CSF SC once daily on days 16-26. Patients also receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 14 days after last GM-CSF injection, patients receive GM-CSF SC once daily on days 1-15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: sargramostim; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Other: laboratory biomarker analysis; Other: immunologic technique

INTERVENTIONS:
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Other: laboratory biomarker analysis — Correlative studies
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological

SUMMARY:
RATIONALE: Colony stimulating factors, such as sargramostim (GM-CSF), may stimulate the immune system in different ways and stop tumor cells from growing and may also increase the number of immune cells found in bone marrow or peripheral blood and help the immune system recover from the side effects of chemotherapy. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving GM-CSF together with paclitaxel albumin-stabilized nanoparticle formulation may be an effective treatment for ovarian cancer, fallopian tube cancer, and primary peritoneal cancer.

PURPOSE: This phase II trial is studying how well giving GM-CSF together with paclitaxel albumin-stabilized nanoparticle formulation works in treating patients with advanced ovarian cancer, fallopian tube cancer, or primary peritoneal cancer that did not respond to previous chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether chronic GM-CSF administration during and after cytotoxic chemotherapy with paclitaxel albumin-stabilized nanoparticle formulation can induce a longer remission than experienced in the most recent platinum-containing regimen.

SECONDARY OBJECTIVES:

I. To determine the extent to which chronic GM-CSF administration can increase the number of activated monocytes in patients with advanced stage epithelial ovarian cancer.

II. To determine the extent to which chronic GM-CSF administration can increase the number and activation state of peripheral circulating antigen presenting cells, such as dendritic cells and activated monocytes, in patients with advanced epithelial ovarian cancer.

III. To determine the extent to which chronic GM-CSF administration can increase the number and functional status of T cells that recognize tumor specific antigens in patients with advanced stage epithelial ovarian cancer.

IV. To determine the extent to which chronic GM-CSF administration can increase the number and functional status of antigen specific T cells that recognize foreign pathogens in patients with advanced stage epithelial ovarian cancer.

OUTLINE:

INDUCTION THERAPY: Patients receive GM-CSF subcutaneously (SC) once daily on days 16-26. Patients also receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Beginning 14 days after last GM-CSF injection, patients receive GM-CSF SC once daily on days 1-15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 6 months and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven epithelial ovarian, fallopian tube or primary peritoneal malignancies, excluding tumors of low malignant potential (borderline)
* Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified
* Patients must have either primary platinum refractory or resistant carcinoma or secondary platinum resistant disease:

  1. Primary platinum refractory disease is defined as progression of disease on initial platinum-based chemotherapy or persistent disease at the conclusion of the initial platinum-based chemotherapy course associated with the primary debulking surgery.
  2. Primary platinum resistant disease is defined as recurrence of carcinoma within 6 months (+ 14 days) of completion of initial platinum-based chemotherapy associated with the primary debulking surgery. (The 14 day window is to allow study entry for those patients where evidence clearly suggests that had an assessment been made early the patient would have met the 6 month time line. This will be determined by the study principal investigator [P.I.])
  3. Secondary platinum resistant disease is defined as meeting any one of the listed criteria during or following a subsequent platinum containing regimen.
* Patients must have an elevated serum cancer antigen (CA)125 on two occasions greater than 7 days apart
* Absolute neutrophil count >= 1500/uL
* Platelets >= 100,000/uL
* Creatinine =< 2.0 mg/dL
* Total bilirubin =< 1.5 mg/dL (unless history of Gilbert's disease)
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 x upper limit of normal (ULN) or < 5 x ULN with documented report of hepatic metastases
* Patients must have recovered from effects of recent surgery, radiotherapy, or chemotherapy; at least three weeks must have elapsed since prior chemotherapy or radiation therapy

Exclusion Criteria:

* Patient has an allergic history to paclitaxel or GM-CSF, not manageable by pre-medication and/or slow drug infusion
* Patient has poorly controlled arrhythmias or unstable coronary artery disease or has had a myocardial infarction within the last six months
* Patient with active pulmonary edema or pleural effusion
* Active infection requiring IV antibiotics
* Patient currently requires lithium, (due to drug interaction with GM-CSF [Leukine])
* Patient currently presents with a neurotoxicity > Grade 1
* Women of childbearing potential
* Patients with a history of other invasive malignancies, within the previous 5 years are excluded, with the exception of non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-05; Primary Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Goff, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Colony Stimulating Factor and Chemotherapy): INDUCTION THERAPY: Patients receive Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) subcutaneously (SC) once daily on days 16-26. Patients also receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 14 days after last GM-CSF injection, patients receive GM-CSF SC once daily on days 1-15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  sargramostim: Given SC
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  laboratory biomarker analysis: Correlative studies
  immunologic technique: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Colony Stimulating Factor and Chemotherapy): INDUCTION THERAPY: Patients receive GM-CSF SC once daily on days 16-26. Patients also receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 14 days after last GM-CSF injection, patients receive GM-CSF SC once daily on days 1-15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  sargramostim: Given SC
  paclitaxel albumin-stabilized nanoparticle formulation: Given IV
  laboratory biomarker analysis: Correlative studies
  immunologic technique: Correlative studies
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Median time to progression
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 21
months | 4.07 [2.74 to 6.71]

2. Primary Outcome: Response Rate
Description: Number of patients achieving a complete or partial response.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 21
Participants | 15

3. Secondary Outcome: Correlation Between Circulating Monocytes and Time to Progression
Description: Baseline median percentages of CD45+ cells made up of monocytes in complete responders (CR) compared to partial-responders, non-responders and those with stable disease (PR+NR+SD).
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: percentage of CD45+ in PBSC
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 21
percentage of CD45+ in PBSC
  CR | 20.75 [10.98 to 24.93]
  PR+NR+SD | 12.75 [11.24 to 30.1]

4. Secondary Outcome: Correlation Between Circulating Dendritic Cell Count and Maturation State With Clinical Response and Response Duration
Description: Baseline median percentages of CD45+ cells made up of myeloid dendritic cells (mDC) and plasmacytoid dendritic cells (pDC) in complete responders (CR) compared to partial and non-responders (PR+NR+SD).
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: % of CD45+PBMC
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 21
% of CD45+PBMC
  mDC in CR | 1.543 [1.075 to 3.504]
  mDC in PR+NR+SD | 1.996 [1.232 to 2.42]
  pDC in CR | 0.2465 [0.1924 to 0.3362]
  pDC in PR+NR+SD | 0.3743 [0.2311 to 0.5067]

5. Secondary Outcome: Precursor Frequency of Circulating Activated T Lymphocytes Against Common Ovarian Cancer Tumor Associated Antigens to Measure the Development of Immunity to Anti-tumor Antigens
Description: Correlation of time to progression and change in circulating activated T lymphocytes from baseline to follow-up.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: Pearson correlation
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 21
Pearson correlation
  IGF1R-p1196-1210 | 0.5056 [-0.03429 to 0.8171]
  IGF1R-p1242-1256 | 0.8496 [0.5807 to 0.9513]
  IGF1R-p1332-1346 | 0.8269 [0.5279 to 0.9435]
  IGFBP2 | 0.3676 [-0.2982 to 0.7927]
  p53 | -0.02268 [-0.5667 to 0.5351]
  PRAME | -0.0817 [-0.5869 to 0.4693]

6. Secondary Outcome: Precursor Frequency of Circulating T Lymphocytes Activated Against Foreign Antigens
Description: Correlation of time to progression and change in circulating activated T lymphocytes from baseline to follow-up.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: Pearson correlation
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Number analyzed (Participants) | 21
Pearson correlation
  PHA | -0.08759 [-0.5908 to 0.4647]
  CEF | -0.1818 [-0.6498 to 0.3862]
  tetanus toxoid | -0.1071 [-0.6035 to 0.4491]

ADVERSE EVENTS:
Arm/Group | Treatment (Colony Stimulating Factor and Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Colony Stimulating Factor and Chemotherapy) (N=21)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Obstruction, GI (Gastrointestinal disorders) | 1 (1)
Abdomen NOS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Colony Stimulating Factor and Chemotherapy) (N=21)
Allergic Reaction/Hypersensitivity (Including drug fever) (Immune system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Low HCT (Blood and lymphatic system disorders) | 2
Hematocrit (Blood and lymphatic system disorders) | 3
RBC (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 13
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 6
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6
Platelets (Blood and lymphatic system disorders) | 2
Hypertension (Cardiac disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Rigors/Chills (General disorders) | 2
Weight Gain (General disorders) | 2
Weight Loss (General disorders) | 2
Death not associated with CTCAE term (General disorders) | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 7
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 6
Nail Changes (Skin and subcutaneous tissue disorders) | 3
Rash: Acne/Acneiform (Skin and subcutaneous tissue disorders) | 2
Anorexia (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 4
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 7
Edema:limb (Blood and lymphatic system disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 2
GFR (Metabolism and nutrition disorders) | 2
Low Protein (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Memory Impairment (General disorders) | 2
Somnolence/depressed level of consciousness (General disorders) | 2
Arthralgia (Pain) (General disorders) | 2
Bone Pain (General disorders) | 4
Head pain/Headache (General disorders) | 4
Joint Pain (General disorders) | 2
Muscle Pain (General disorders) | 3
Myalgia (Pain) (General disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Urinary Retention (including neurogenic bladder) (Renal and urinary disorders) | 2
Flu-like syndrome (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes